CLINICAL TRIAL: NCT07403968
Title: An Open-Label, Single-Arm, Phase 2a Trial to Evaluate the Safety, Tolerability, PK, and Mechanism of Action of Zasocitinib (TAK-279) in Participants With Active Crohn's Disease
Brief Title: A Study of Zasocitinib (TAK-279) in Adults With Active Crohn's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-279-CD-2003
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zasocitinib Dose (Experimental): Participants will receive zasocitinib dose orally, once daily (QD) for 12 week treatment period (Week 0 to 12).
  Interventions: Drug: Zasocitinib

INTERVENTIONS:
Drug: Zasocitinib — Zasocitinib administered orally.
  Other Names: TAK-279

SUMMARY:
Crohn's disease (CD) is a serious, long-term condition that can cause swelling (inflammation) and painful ulcers anywhere in the gut. The main aim of this study is to evaluate how safe zasocitinib is and how well it is tolerated by adults with CD.

The participants will be treated with zasocitinib for 3 months (12 weeks) and will need to undergo a test where a doctor uses a thin, flexible tube with a tiny camera to look inside the large bowel (colon) and the end of the small bowel (ileum); this test is called ileocolonoscopy.

During the study, participants will visit the study clinic several times.

DETAILED DESCRIPTION:
The drug being tested in this study is zasocitinib. Zasocitinib is being tested to treat participants with active Crohn's disease. The study will look at the safety of zasocitinib.

The study will enroll approximately 20 participants. This is a single center study. The overall duration is up to approximately 5 months (20 weeks) including a 4-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 75 years can participate in the study.
2. Must have been diagnosed with Crohn's disease (CD) at least 1 month (30 days) before study start.
3. Must have received other treatments for CD earlier but no longer tolerate these treatments or the treatment no longer helps.

Exclusion Criteria

1. Cannot have another condition that causes swelling (inflammation) in the bowel.
2. Cannot have complications of CD which may require surgery.
3. Cannot have current abscesses or abscesses that have been treated within 6 weeks before study start.
4. Cannot have had a removal of parts of the bowel within half a year (6 months) before study start.
5. Cannot have had any surgery inside the belly (intraabdominal) within 3 months before study start.
6. Cannot have or had a J-pouch.
7. Cannot have had infections up to 2 months (8 weeks) before study start.
8. Cannot have given blood or plasma within 1 month (30 days) before study start.
9. Cannot tolerate having blood taken with a needle from a vein (venipuncture).

Additional entry criteria will be discussed with the study doctor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-05-16 (Estimated); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) and Adverse Events of Special Interests (AESIs) | From start of study drug administration up to follow-up (up to Week 16)
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the trial intervention, whether or not the occurrence is considered related to the trial intervention. A TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a trial intervention or medicinal product or any existing event that worsens in either intensity or frequency after exposure to the trial intervention. An AESI is an adverse event of scientific and medical concern specific to the compound or program, for which ongoing monitoring and rapid communication by the investigator may be appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/